CLINICAL TRIAL: NCT03243617
Title: A Placebo-Controlled, Double-Blind, Bi-Lateral Study to Evaluate the Performance and Tolerability of a Cosmetic Product Designed to Improve the Appearance of Skin Afflicted With Keratosis Pilaris
Brief Title: Cosmetic Study of AO+Mist in Improving the Appearance of Skin Afflicted With Keratosis Pilaris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AOBiome LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AOB2015-02
Record Dates: First submitted 2017-08-01; First posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Keratosis Pilaris
MeSH Terms: conditions — Burnett Schwartz Berberian syndrome

STUDY DESIGN:
Intervention Model Description: Bi-Lateral study
Who Masked: Participant, Care Provider
Masking Description: AO+ Mist (or placebo) are supplied in white 100mL metered spray bottles. Test products are blinded and labeled for application to the LEFT or RIGHT side of the body.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AO+Mist (Active Comparator): Cosmetic Product AO+Mist
  Interventions: Other: Placebo; Other: AO+Mist
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo; Other: AO+Mist

INTERVENTIONS:
Other: Placebo — Subjects are instructed in the use of the spray bottle and asked to self-administer the Test Product as follows:
  * LEFT side of the body where skin is affected: Five (5) pumps of Spray (BOTTLE LABELED: LEFT) must be applied twice-a-day to the entire area affected by KP once in the morning and once in the evening for 28 days.
  * RIGHT side of the body where skin is affected: Five (5) pumps of Spray (BOTTLE LABELED: RIGHT) must be applied twice-a-day to the entire area affected by KP once in the morning and once in the evening for 28 days.
  * Subjects may not wash their body with soap and water AFTER the applications
Other: AO+Mist — Subjects are instructed in the use of the spray bottle and asked to self-administer the Test Product as follows:
  * LEFT side of the body where skin is affected: Five (5) pumps of Spray (BOTTLE LABELED: LEFT) must be applied twice-a-day to the entire area affected by KP once in the morning and once in the evening for 28 days.
  * RIGHT side of the body where skin is affected: Five (5) pumps of Spray (BOTTLE LABELED: RIGHT) must be applied twice-a-day to the entire area affected by KP once in the morning and once in the evening for 28 days.
  * Subjects may not wash their body with soap and water AFTER the applications

SUMMARY:
The purpose of this study is to demonstrate the safety, tolerability and efficacy of AO+ Mist administered daily for 4 weeks to improve the appearance of skin afflicted with keratosis pilaris.

DETAILED DESCRIPTION:
This will be a single center, double-blind, placebo-controlled study in subjects with keratosis pilaris affecting both sides of the body.

Subjects will be screened within 4 weeks of enrollment. Subjects will be seen at the research facility on for the baseline visit and will be asked to return to the site on weeks 1, 2, 3 and 4 for assessments. Test product application will occur for four weeks starting with the day of the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects ≥18 and ≤65 years of age
2. Subject is in good general health
3. Diagnosis of keratosis pilaris involving areas of the body affected bilaterally
4. Subject has Fitzpatrick Skin Type I-VI
5. Willing to refrain from using any treatments, other than the investigational product, including antibiotics, for acne present on the face.
6. Ability to comprehend and comply with procedures
7. Agree to commit to participate in the current protocol
8. Provide written informed consent prior to any study procedure being performed (all subjects should be able to understand the informed consent form and any other documents that subjects are required to read)

Exclusion Criteria:

1. Male and female subjects under 18 years or over 65 years of age
2. Female subjects who are pregnant or lactating
3. Subjects who have received laser therapy to the KP affected area in the past 1 year
4. Subjects with a concurrent diagnosis of another skin condition or malignancy
5. Subjects with tan or sunburn over the area affected by KPin the past month
6. Subjects with open, non-healing sores or infections at any skin site
7. Treatment with over-the-counter topical medications for the treatment of acne vulgaris including benzoyl peroxide, topical anti-inflammatory medications, corticosteroids, α-hydroxy/glycolic acid, including lactic acid lotions (Am-Lactin, Lac-Hydrin), urea cream (Carmol 10, Carmol 20, Carmol 40, Urix 40), salicylic acid (Salex lotion), topical corticosteroids within 4 weeks prior to baseline.
8. Treatment with systemic corticosteroids (including intranasal and inhaled corticosteroids) within 4 weeks prior to baseline
9. Treatment with systemic antibiotics or systemic anti-acne drugs or systemic anti-inflammatory drugs within 4 weeks prior to baseline
10. Prescription topical retinoid use on the face or body within 4 weeks of baseline (e.g., tretinoin, tazarotene, adapalene).
11. Oral retinoid use (e.g., isotretinoin) within 12 months prior to baseline or vitamin A supplements greater than 10,000 units/day within 6 months of baseline..
12. Treatment with any investigational drug within 30 days prior to the beginning of the screening period (this includes investigational formulations of marketed products, inhaled and topical drugs)
13. Subjects who are unable to understand the protocol or give informed consent
14. Any other condition and/or situation that causes the Investigator to deem a subject unsuitable for the study (e.g., due to expected study medication non-compliance, inability to medically tolerate the study procedures, or a subject's unwillingness to comply with study-related procedures)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-12-04 (Actual); Primary Completion 2016-06-08 (Actual); Study Completion 2016-09-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as assessed by physical exam and appearance | Baseline-Week 4

SECONDARY OUTCOMES:
Difference in Keratosis pilaris Investigator Score | Baseline-Week 4

OTHER OUTCOMES:
Difference in Skindex16 Quality of Life survey | Baseline-Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Dover, MD, Principal Investigator — Skincare Physicians
Locations (1):
- Skincare Physicians, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No